CLINICAL TRIAL: NCT05401383
Title: Implementation of Upper Gi Endoscopy Preparation: RCT Fasting Versus Lumevis
Brief Title: Implementation of Upper Gi Endoscopy Preparation: Fasting Versus Lumevis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Azienda USL Modena (Other)
Responsible Party: Principal Investigator, Dr. Mauro Manno, Director of Gastroenterology and Digestive Endoscopy Unit, Azienda USL Modena
Other Study IDs: AziendaUSLModena
Record Dates: First submitted 2022-05-27; First posted 2022-06-02 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2022-05

CONDITIONS: EGDS Preparation; Fasting; Lumevis
MeSH Terms: conditions — Fasting

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: fasting from solids (6 hours before) and clear fluids (2 hours before the exam)
- Group B: Lumevis intake (50 ml), 30 minutes before the exam plus fasting as group A
  Interventions: Device: Lumevis (IIa class)

INTERVENTIONS:
Device: Lumevis (IIa class) — intake of Lumevis 30 minutes before EGDS
  Groups: Group B

SUMMARY:
One of the major problems for the endoscopist during esophagogastroduodenoscopy (EGDS) is the presence of foam, bubbles, mucus and saliva, whether small or large, which can compromise correct endoscopic visibility. Endoscopy of the upper gastrointestinal tract, like that of the lower gastrointestinal tract, requires optimal visualization of the mucosa. It is clear that endoscopic vision is often hindered by the presence of bubbles and foam: multiple aspirations alternating with intraprocedural washes are therefore necessary, which lengthen the time necessary for the endoscopic examination. Nowadays there's no universal raccomandation about a specific preparation before EGDS.

The aim of our study is to compare fasting versus the use of simethicone premedication in combination with N-acetyl- cysteine and acetic acid (LumevisTM).

The study is observational, randomized 1:1, and double blind. Primary outcomes are: grade of mucosa visualization defined by visual analogue scale (0-10) for each analyzed segment (esophagus, stomach and duodenum).

Secondary aims: general patient satisfaction defined by visual analogue scale, eventual adverse events, duration of the exam.

ELIGIBILITY:
Inclusion Criteria:

* adult patients that underwent EGDS

Exclusion Criteria:

* previous upper GI surgery
* previous endoscopic bariatric procedures
* known upper GI stenosis (benign and malign)
* previous diagnosis of achalasia or motility disorders
* diabetes
* allergy to one of lumevis components
* cystinuria
* fasting not correctly respected
* pregnant or brest-feeding women
* urgent-emercengy setting
* inpatients
* patients who don't give their consent to partecipate to the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: adult patients who had to perform EGDS
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
grade of mucosa visibility | 6 months
  evalueted by VAS after the exam (it will be recorded a video) by a physician that not performed the exam and that are blinded about the randomization

SECONDARY OUTCOMES:
general patient satisfaction | 6 months
  evalueted by VAS at the end of the exam, before the discharge to home
eventual adverse events | 6 months
  evalueted by ASGE lexicon, at the end of the exam, before the discharge to home
duration of the exam | 6 months
  minutes between intubation and extubation of the endoscope from the mouth

CONTACTS AND LOCATIONS:
Locations (1):
- Mauro Manno, Carpi, MO, Italy

IPD SHARING:
Plan to Share IPD: No